CLINICAL TRIAL: NCT03397303
Title: Quantification of Nerve Stiffness in Patients with Peripheral Neuropathies
Brief Title: Quantification of Nerve Stiffness in Neuropathies
Acronym: Nerf_SSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Université de Nantes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RC17_0231
Record Dates: First submitted 2018-01-05; First posted 2018-01-11 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy; Charcot-Marie-Tooth Disease, Type IA; Anti-MAG Neuropathy
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Charcot-Marie-Tooth Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- patients with peripheral neuropathies (Experimental): This project aims to understand how nerve mechanical properties are altered in patients with rare peripheral neuropathies . Stiffness of various peripheral nerves will be measured using ultrasound shear wave elastography. Patients will be compared with age-matched controls.
  Interventions: Other: elastography measurements
- controls (Other)
  Interventions: Other: elastography measurements

INTERVENTIONS:
Other: elastography measurements — elastography measurements

SUMMARY:
This project aims to understand how nerve mechanical properties are altered in patients with rare peripheral neuropathies . Stiffness of various peripheral nerves will be measured using ultrasound shear wave elastography. Patients will be compared with age-matched controls.

DETAILED DESCRIPTION:
The following nerve will be studied bilaterally, in a randomised order: Median, ulnar, Radial, Sciatic and Tibial.

Participants will be asked to remain relaxed during elastography measurements.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 65
* Having social insurance status
* Having given informed consent
* Diagnostic of chronic inflammatory demyelinating polyradiculoneuropathy (CIDP), CMT1a or Anti-MAG (peak immunoglobulin M (IGm)>15,000 BTU)

Exclusion Criteria:

For controls:

* Person staying in a health or social facility
* Person unable to understand the protocol and to respect the modalities
* Person deprived of liberty
* Person of legal age benefiting from a system of legal protection (guardianship, curators or safeguard of justice)
* Participation in another biomedical research in progress
* Diabetes, history of neuromuscular disease

For CIDP:

* Person staying in a health or social facility
* Person unable to understand the protocol and to respect the modalities
* Person deprived of liberty
* Person of legal age benefiting from a system of legal protection (guardianship, curators or safeguard of justice)
* Participation in another biomedical research in progress
* MRC score < 3

For Charcot-Marie-Tooth type 1 (CMT1) and anti-MAG:

* Person staying in a health or social facility
* Person unable to understand the protocol and to respect the modalities
* Person deprived of liberty
* Person of legal age benefiting from a system of legal protection (guardianship, curators or safeguard of justice)
* Participation in another biomedical research in progress

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2023-12-08 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
nerve shear wave velocity | Day0
  Ultrasound shear wave elastography will provide a measure of nerve shear wave velocity, which will be used as a surrogate of nerve stiffness.

CONTACTS AND LOCATIONS:
Overall Officials: Yann Pereon, PU-PH, Principal Investigator — Nantes University Hospital
Locations (1):
- Univeristy of Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: No